CLINICAL TRIAL: NCT04827264
Title: Safe Return to Play Following ACL Reconstruction: Validation of a Return to Play Checklist
Brief Title: Safe Return to Play After ACL Reconstruction
Status: Completed | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: KFREE16D.026
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Return to Play Testing using Checklist: Participants will be evaluated prospectively for return to play following ACL reconstruction by testing with the "Safe return to play following ACL reconstruction checklist"
  Interventions: Diagnostic Test: Safe Return to Play Following ACL Reconstruction Checklist
- Return to Play Testing using Clinical Judgment: Participants will be evaluated prospectively for return to play following ACL reconstruction by testing with clinical judgement

INTERVENTIONS:
Diagnostic Test: Safe Return to Play Following ACL Reconstruction Checklist — All participants who have undergone primary ACL reconstruction will receive PT evaluation using our "Return to Play Checklist" at 7 months post-op, prior to return to sports
  Groups: Return to Play Testing using Checklist

SUMMARY:
Recent studies report that as few as 44% of athletes undergoing ACL reconstruction were able to return to their prior level of competitive level of sports. Early return may predispose an individual to re-injury including graft re-tear, meniscal tears, chondral injuries, and contralateral knee injuries. Criteria governing clearance to return to sports after ACL reconstruction has been traditionally defined using time from surgery and one or two objective criteria, often solely isokinetic quad/hamstring strength. Several studies have suggested that historical criteria used to assess readiness to return to play (RTP) are insufficient in identifying individuals at risk of a re-injury. They advocate for additional functional and dynamic testing, which may better reflect the complex kinematics required in high level athletic competition.

We previously developed a "Safe Return to Play Following ACL Reconstruction Checklist" based on a systematic review of the literature and expert survey. Seven objective measures were developed as part of the checklist. The checklist is performed by a certified physical therapist trained in these performance tests.

The purpose of this study is to validate the utility of our "Return to Play Checklist" by evaluating our patients prospectively for return to play following ACL reconstruction by comparing a cohort of patient undergoing testing with the checklist versus "clinical judgement."

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 15-35 undergoing primary ACL reconstruction

Exclusion Criteria:

* patients who are undergoing revision ACL surgery

Ages: 15 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants ages 15-35 who have undergone primary ACL reconstruction at Rothman Orthopaedics
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2016-02-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Return to Play | 7 months
  Participants will be evaluated prior to returning to sports using the "return to play checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States